CLINICAL TRIAL: NCT05303818
Title: Evaluation of Chemoprophylaxis With Rivaroxaban for Lower Limb Deep Vein Thrombosis in the Surgical Treatment of Colorectal Cancer
Brief Title: Chemoprophylaxis With Rivaroxaban for Lower Limb Deep Vein Thrombosis in Colorectal Cancer
Acronym: Ésquilo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, Rafael de Athayde Soares, PhD, MsC, M.D - Investigador Principal - médico preceptor do Serviço de Cirurgia Vascular, Hospital do Servidor Publico Estadual
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 34953614.3.0000.5463
Record Dates: First submitted 2022-02-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Deep Venous Thrombosis; Colonic Cancer
Keywords: deep vein thrombosis,; colonic cancer
MeSH Terms: conditions — Venous Thrombosis; Colonic Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: 68 patients will be selected for the study. All patients must complete an informed consent form regarding the objectives and risks involved in this research
Masking Description: Patients information will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- post-operative patients with colonic cancer (Experimental): Patients will receive Rivaroxaban 10mg/daily for 28 days after surgery. Only one arm.
  Interventions: Drug: Rivaroxaban 10 MG

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Patients in post-operative colonic cancer will receive rivaroxaban 10mg/daily for 28 days after surgery

SUMMARY:
The chemoprophylaxis of deep vein thrombosis (DVT) with subcutaneous low-molecular-weight heparin (enoxaparin) in the postoperative period of elective surgeries is already well established in the literature and in clinical practice. However, the use of this medication can have a financial impact on the patient and the parenteral presentation itself is associated with pain at the application site, which can make it difficult for patients to adhere.

DETAILED DESCRIPTION:
There are already robust studies in the literature demonstrating the efficacy and safety of using Rivaroxaban 10mg once a day in the prevention of deep vein thrombosis of the lower limbs in patients undergoing orthopedic knee and hip surgeries.1,2,3 Although there are already trials demonstrating the safety and efficacy of the use of rivaroxaban in the treatment of DVT and venous thromboembolism in cancer patients, there is a lack in the literature, to date, of studies on the efficacy and safety of prophylaxis with Ribaroxaban for DVT of the lower limbs in the post-operative period. operative of colorectal cancer surgeries, both open surgeries and videolaparoscopic surgeries.4 There are robust studies in the literature, with about 3645 patients undergoing colorectal cancer surgery, reporting a VTE incidence of about 0.85%. .OBJECTIVE To determine the efficacy and safety of chemoprophylaxis for DVT with Rivaroxaban in patients undergoing surgical treatment of colorectal cancer. Primary objective: prevention of DVT and VTE in patients after colorectal surgery. Secondary objective: rates of bleeding and adverse events in patients undergoing anticoagulant use.

METHOD This is a prospective, observational cohort of patients undergoing surgical treatment for colorectal cancer at the Digestive System and Coloproctology Surgery service at Hospital do Servidor Público Estadual de São Paulo. Patients undergoing chemoprophylaxis with enoxaparin and rivaroxaban to prevent lower limb DVT after surgical treatment of colorectal cancer will be included.

In the immediate postoperative period, they will be submitted to chemoprophylaxis with Enoxaparin 40mg subcutaneously 1x/day for 24 hours up to a maximum of 7 days, depending on the release of the diet and the need for a new surgical approach, and at hospital discharge, Rivaroxaban 10mg orally 1x/day will be prescribed until complete 28 days of prophylactic anticoagulation after surgery. Before surgery and after the last dose of chemoprophylaxis, patients will be evaluated with venous USG-Doppler of the lower limbs, in order to detect any possibility of asymptomatic deep vein thrombosis. In addition, 1 week after hospital discharge, patients will be evaluated for symptoms related to the lower limbs in a return visit, as well as any bleeding resulting from the use of drugs for DVT chemoprophylaxis (Table 1).

For the diagnosis of DVT we will use clinical and laboratory data and especially venous Doppler ultrasound. The main ultrasound data used for the diagnosis of DVT are vessel incompressibility and lack of flow in the analyzed vessels.5,6 Venous Doppler US will be performed by an examiner blinded to the treatment received by the patient, with compression measurements in the common femoral veins, superficial in the middle third and popliteal vein. The evaluation of venous recanalization will be through verification of total, partial or absent venous flow. In addition, the presence of venous reflux and its degree will be quantified.

Diagnostic criteria for acute DVT on Doppler: absence or decrease in venous compression; visible thrombus; increase in venous diameter; no increase in venous diameter with Valsalva; valve immobility; loss of respiratory phasicity; absence or decrease in spontaneous venous flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients in post-operative surgery for colonic cancer.
* No contraindication for anticoagulation usage.
* Absence of renal or hepatic failure.

Exclusion Criteria:

* Pregnancy,
* age < 18 years,
* contraindication to the use of anticoagulants, -failure to complete the informed consent form. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Deep venous thrombosis and embolic pulmonary disease | 28 days after surgery
  Patients will evaluated with Duplex ultrasound. Duplex ultrasound using b mode and compressibility. All patients will be evaluated.

SECONDARY OUTCOMES:
Safety of rivaroxaban | 28 days after surgery
  Patients will evaluated with Duplex ultrasound. Duplex ultrasound using b mode and compressibility. All patients will be evaluated. Safety will be evaluated regarding bleeding and no thrombosis afterall.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Servidor Público Estadual de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plan to share data.